CLINICAL TRIAL: NCT01068912
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Multicenter Study Evaluating the Efficacy and Safety of Two Doses of Favipiravir in Adult Patients With Uncomplicated Influenza
Brief Title: Dose-Finding Study of Favipiravir in the Treatment of Uncomplicated Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MDVI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T705aUS204
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1: Experimental (Experimental): Low-dose favipiravir regimen: 1000 mg favipiravir twice a day (BID) x 1 day, and 400 mg favipiravir BID x 4 days
  Interventions: Drug: Favipiravir
- 2: Experimental (Experimental): High-dose favipiravir regimen: 1200 mg favipiravir BID x 1 day, and 800 mg favipiravir BID x 4 days
  Interventions: Drug: Favipiravir
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Favipiravir — 1000 mg favipiravir BID x 1 day, and 400 mg favipiravir BID x 4 days
  Arms: 1: Experimental
Drug: Favipiravir — High-dose favipiravir regimen: 1200 mg favipiravir BID x 1 day, and 800 mg favipiravir BID x 4 days
  Arms: 2: Experimental
Drug: Placebo comparator — Placebo BID x 1 day, and Placebo BID x 4 days
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled multicenter study evaluating the efficacy and safety of two doses of favipiravir in adult patients with uncomplicated influenza.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study designed to evaluate the efficacy and safety of a 5-day regimen of favipiravir in influenza patients aged 20-80 years. Enrolled patients will be randomly assigned to 1 of 3 parallel treatment dose groups:Placebo; Low-dose favipiravir (1000 mg favipiravir BID for 1 day, followed by 400 mg favipiravir BID for 4 days); High-dose favipiravir (1200 mg favipiravir BID for 1 day, followed by 800 mg favipiravir BID for 4 days).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who test positive for influenza A or B by a commercially available Rapid Antigen Test (RAT) of the nasopharynx. A patient with a negative RAT result may still enroll if the sponsor and investigator agree that there is a known influenza outbreak circulating in the community.
2. Patients ≥ 20 but < 65 years of age with a temperature (oral) of 100.4°F (38.0°C) or more; patients ≥ 65 years of age with a temperature (oral) of 100.0°F (37.8°C) or more at the first visit, or in the 6 hours prior if antipyretics were taken.
3. Patients with 2 or more of the following symptoms (moderate to severe in intensity) at the time of enrollment:

   * Cough
   * Sore throat
   * Headache
   * Nasal congestion
   * Feeling feverish
   * Body aches and pains
   * Fatigue (tiredness)

Exclusion Criteria:

1. Patients who have had influenza symptoms or fever (i.e., one of the symptoms listed under the inclusion criteria) for 36 hours or more prior to study screening.
2. Patients who have underlying chronic respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], chronic bronchitis, diffuse panbronchiolitis, bronchiectasis, pulmonary emphysema, pulmonary fibrosis, bronchial asthma, or old tuberculosis).
3. Patients who at the beginning of the study are suspected of having bacterial respiratory infection (i.e., expectoration of purulent or mucopurulent sputum and/or infiltrate in lung in a chest x-ray, etc.).
4. Patients who have serious chronic diseases. For example, patients with HIV, cancer (i.e., requiring chemotherapy within the preceding 6 months), cirrhosis (end-stage), and/or unstable renal, cardiac, pulmonary, neurologic, vascular, or endocrinologic disease states requiring medication dose adjustments within the last 30 days.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Macy Guiont, Study Director — Syneos Health
Locations (228):
- United States (148):
  - #065, Birmingham, Alabama
  - #156, Huntsville, Alabama
  - #151, Mobile, Alabama
  - #155, Scottsboro, Alabama
  - #173, Toney, Alabama
  - #161, Tuscumbia, Alabama
  - #089, Chandler, Arizona
  - #018, Green Valley, Arizona
  - #110, Mesa, Arizona
  - #105, Phoenix, Arizona
  - #188, Tucson, Arizona
  - #107, Jonesboro, Arkansas
  - #019, North Little Rock, Arkansas
  - #140, Searcy, Arkansas
  - #059, Anaheim, California
  - #179, Anaheim, California
  - #032, Chino, California
  - #154, Cypress, California
  - #004, Garden Grove, California
  - #144, Long Beach, California
  - #043, Los Angeles, California
  - #139, Los Angeles, California
  - #096, Oxnard, California
  - #091, Pacific Palisades, California
  - #114, Pasadena, California
  - #111, Pico Rivera, California
  - #097, Pomona, California
  - #068, Sacramento, California
  - #035, San Diego, California
  - #054, San Diego, California
  - #042, Torrance, California
  - #197, Bridgeport, Connecticut
  - #022, Boca Raton, Florida
  - #152, Boynton Beach, Florida
  - #060, Coral Gables, Florida
  - #007, Delray Beach, Florida
  - #086, Edgewater, Florida
  - #016, Fort Myers, Florida
  - #038, Gainesville, Florida
  - #014, Hialeah, Florida
  - #052, Hialeah, Florida
  - #088, Hialeah, Florida
  - #035, Jacksonville, Florida
  - #094, Kissimmee, Florida
  - #153, Kissimmee, Florida
  - #177, Lauderdale Lakes, Florida
  - #012, Melbourne, Florida
  - #034, Miami, Florida
  - #040, Miami, Florida
  - #047, Miami, Florida
  - #082, Miami, Florida
  - #166, Miami, Florida
  - #149, Miami Gardens, Florida
  - #134, Pinellas Park, Florida
  - #050, Port Orange, Florida
  - #163, Venice, Florida
  - #020, West Palm Beach, Florida
  - #814, Snellville, Georgia
  - #080, Honolulu, Hawaii
  - #063, Boise, Idaho
  - #835, Oak Lawn, Illinois
  - #804, Fishers, Indiana
  - #803, Franklin, Indiana
  - #198, Greenfield, Indiana
  - #195, Munci, Indiana
  - #168, Council Bluffs, Iowa
  - #827, West Des Moines, Iowa
  - #008, Newton, Kansas
  - #138, Shawnee, Kansas
  - #106, Wichita, Kansas
  - #055, Hazard, Kentucky
  - #823, Alexandria, Louisiana
  - #801, Baton Rouge, Louisiana
  - #048, Elkridge, Maryland
  - #085, Silver Spring, Maryland
  - #187, Worcester, Massachusetts
  - #811, Detroit, Michigan
  - #015, Bellevue, Nebraska
  - #170, Bellevue, Nebraska
  - #081, Lincoln, Nebraska
  - #017, Omaha, Nebraska
  - #041, Omaha, Nebraska
  - #169, Omaha, Nebraska
  - #112, Henderson, Nevada
  - #146, Henderson, Nevada
  - #079, Las Vegas, Nevada
  - #176, Las Vegas, Nevada
  - #171, Brooklyn, New York
  - #011, Endwell, New York
  - #164, New York, New York
  - #021, Harrisburg, North Carolina
  - #178, High Point, North Carolina
  - #189, Morganton, North Carolina
  - #030, Carlisle, Ohio
  - #006, Cleveland, Ohio
  - #182, Grove City, Ohio
  - #083, Wadsworth, Ohio
  - #167, Oklahoma City, Oklahoma
  - #810, Oklahoma City, Oklahoma
  - #071, Tulsa, Oklahoma
  - #045, Portland, Oregon
  - #024, Bridgeville, Pennsylvania
  - #815, Clairton, Pennsylvania
  - #192, Harleysville, Pennsylvania
  - #816, Philladelphia, Pennsylvania
  - #191, Pittsburgh, Pennsylvania
  - #828, Scottdale, Pennsylvania
  - #824, Uniontown, Pennsylvania
  - #194, Johnston, Rhode Island
  - #819, Clinton, South Carolina
  - #805, Easley, South Carolina
  - #160, Murrells Inlet, South Carolina
  - #833, Orangeburg, South Carolina
  - #831, Pawleys Island, South Carolina
  - #147, Simpsonville, South Carolina
  - #002, Rapid City, South Dakota
  - #084, Clarksville, Tennessee
  - #001, Amarillo, Texas
  - #812, Arlington, Texas
  - #137, Austin, Texas
  - #037, Beaumont, Texas
  - #113, Bryan, Texas
  - #058, Carrollton, Texas
  - #066, Corpus Christi, Texas
  - #039, Houston, Texas
  - #053, Houston, Texas
  - #132, Houston, Texas
  - #136, Houston, Texas
  - #157, Houston, Texas
  - #158, Katy, Texas
  - #003, San Antonio, Texas
  - #108, San Antonio, Texas
  - #180, San Antonio, Texas
  - #817, San Antonio, Texas
  - #818, San Antonio, Texas
  - #830, Sugar Land, Texas
  - #135, Tomball, Texas
  - #809, Tomball, Texas
  - #822, Draper, Utah
  - #090, Orem, Utah
  - #117, Salt Lake City, Utah
  - #832, Salt Lake City, Utah
  - #825, South Jordan, Utah
  - #133, West Jordan, Utah
  - #142, Alexandria, Virginia
  - #800, Alexandria, Virginia
  - #009, Richmond, Virginia
  - #172, Spokane, Washington
- Australia (18):
  - #216, Blacktown, New South Wales
  - #207, Burwood, New South Wales
  - #214, Carlton, New South Wales
  - #208, Darlinghurst, New South Wales
  - #205, Glebe, New South Wales
  - #201, Maroubra, New South Wales
  - #218, Neutral Bay, New South Wales
  - #202, Sydney, New South Wales
  - #204, Sydney, New South Wales
  - #219, Biggera Waters, Queensland
  - #215, Caboolture, Queensland
  - #221, Deception Bay, Queensland
  - #217, Jimboomba, Queensland
  - #220, Nerang, Queensland
  - #206, Sherwood, Queensland
  - #223, Mirrabooka, Western Australia
  - #222, Morley, Western Australia
  - #224, Spearwood, Western Australia
- Chile (12):
  - #613, Antofagasta
  - #612, Curicó
  - #606, Quillota
  - #614, Rancagua
  - #603, Santiago
  - #607, Santiago
  - #609, Santiago
  - #610, Santiago
  - #602, Talca
  - #600, Temuco
  - #601, Temuco
  - #611, Viña del Mar
- New Zealand (7):
  - #306, Otara, Auckland
  - #305, Rotorua, Bay of Plenty
  - #302, Tauranga, Bay of Plenty
  - #301, Christchurch, Canterbury
  - #304, Dunedin, Otago
  - #307, Auckland
  - #308, Hamilton
- Paraguay (4):
  - #703, Esquina Pai Perez, Asunción
  - #702, Florida, Asunción
  - #707, Pai Perez, Asunción
  - #704, Campos Cervera, Luque
- Peru (17):
  - #505, Arequipa
  - #511, Callao
  - #506, Cusco
  - #513, Ica
  - #500, Lima
  - #501, Lima
  - #502, Lima
  - #504, Lima
  - #508, Lima
  - #509, Lima
  - #510, Lima
  - #512, Lima
  - #515, Lima
  - #516, Lima
  - #517, Lima
  - #514, Piura
  - #507, Trujillo
- South Africa (22):
  - #421, Benoni
  - #402, Cape Town
  - #405, Durban
  - #406, Durban
  - #408, Durban
  - #412, Durban
  - #414, Durban
  - #404, Johannesburg
  - #422, Kempton Park
  - #411, Kraaifontein
  - #410, Krugersdorp
  - #407, Port Elizabeth
  - #409, Pretoria
  - #413, Pretoria
  - #415, Pretoria
  - #418, Pretoria
  - #419, Pretoria
  - #420, Pretoria
  - #423, Pretoria
  - #417, Sandton
  - #416, Somerset West
  - #401, Soweto

REFERENCES:
- [Derived] Hayden FG, Lenk RP, Epstein C, Kang LL. Oral Favipiravir Exposure and Pharmacodynamic Effects in Adult Outpatients With Acute Influenza. J Infect Dis. 2024 Aug 16;230(2):e395-e404. doi: 10.1093/infdis/jiad409. PMID 37739792

RESULTS

PARTICIPANT FLOW:
Groups:
- 1: Low Dose Favipiravir: Favipiravir: 1000 mg favipiravir BID x 1 day, and 400 mg favipiravir BID x 4 days
- 2: High Dose Favipiravir: Favipiravir: 1200 mg favipiravir BID x 1 day, and 800 mg favipiravir BID x 4 days
Period: Overall Study
Arm/Group | 1: Low Dose Favipiravir | 2: High Dose Favipiravir | Placebo
Started | 134 | 195 | 201
Completed | 123 | 173 | 186
Not Completed | 11 | 22 | 15
Not completed — Adverse Event | 2 | 3 | 2
Not completed — Withdrawal by Subject | 5 | 6 | 6
Not completed — Lost to Follow-up | 3 | 7 | 3
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — aggravation influenza | 1 | 1 | 1
Not completed — other underlying illness | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: The Safety Population, defined as all patients who received study drug, was used for demographic and baseline characteristics and safety analyses, unless otherwise indicated.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Low Dose Favipiravir | 2: High Dose Favipiravir | Placebo | Total
Number analyzed (Participants) | 132 | 189 | 197 | 518
Age, Continuous [Mean (Full Range); unit: years] | 42.2 [20 to 79] | 42.6 [20 to 75] | 42.7 [20 to 80] | 42.5 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 102 | 109 | 284
  Male | 59 | 87 | 88 | 234
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 7 | 4 | 14
  Black or African American | 17 | 22 | 23 | 62
  Hispanic or Latino | 15 | 25 | 29 | 69
  Mestizo | 14 | 20 | 17 | 51
  Native Hawaiian or other Pacific Islander | 2 | 2 | 1 | 5
  White | 72 | 103 | 115 | 290
  Other | 7 | 7 | 6 | 20
  More than one race, including Hispanic or Latino | 0 | 3 | 2 | 5
  More than one race, excluding Hispanic or Latino | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 85 | 120 | 128 | 333
  Peru | 24 | 36 | 36 | 96
  Australia | 7 | 9 | 8 | 24
  South Africa | 8 | 10 | 8 | 26
  Chile | 2 | 9 | 7 | 18
  New Zealand | 6 | 5 | 10 | 21
Rapid Antigen Test Result [Number; unit: participants] — Tested positive for influenza A or B by a commercially available rapid antigen test of the nasopharynx. A patient with a negative rapid antigen test result was enrolled if the sponsor and investigator agreed that there was a known influenza outbreak circulating in the community.
  participants
    Type A Positive | 77 | 113 | 124 | 314
    Type B positive | 30 | 45 | 43 | 118
    Type A and B positive | 6 | 5 | 2 | 13
    Influenza negative | 19 | 26 | 28 | 73
Virus type identification [Number; unit: participants]
  A (H1N1) pdm | 39 | 32 | 39 | 110
  A (H3N2) | 29 | 67 | 66 | 162
  B | 20 | 23 | 20 | 63
  Other | 1 | 0 | 0 | 1
  Neither | 43 | 67 | 72 | 182

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy of 2 Dose Regimens of Favipiravir Compared With Placebo in Treating Patients With Influenza
Description: Overall time required from first study drug administration to alleviation of the 6 primary influenza symptoms and for temperature (oral) measurements to be less than 38.0°C for patients aged 20 to less than 65 years and less than 37.8°C for patients aged 65 years or older. "Alleviated" was defined as all 6 symptom scores had to be decreased to 1 or below and the decrease remain unchanged for 21.5 hours.
Time Frame: 22 weeks
Population: The primary analysis population for efficacy analyses was the ITTI Population (N=333), defined as all patients who received at least 1 dose of study drug with any available efficacy data after randomization and who tested positive for influenza A or B by PCR assay or culture tests on Day 1 using determinations.
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- 2: High Dose Favipiravir: Favipiravir:1200 mg favipiravir BID x 1 day, and 800 mg favipiravir BID x 4 days
Arm/Group | 1: Low Dose Favipiravir | 2: High Dose Favipiravir | Placebo
Number analyzed (Participants) | 88 | 121 | 124
hours | 100.4 [82.4 to 119.8] | 86.5 [79.2 to 102.1] | 91.9 [70.3 to 105.4]
Statistical Analysis 1: Comparison: 1: Low Dose Favipiravir vs 2: High Dose Favipiravir vs Placebo; Time required from first study drug administration to alleviation of the 6 primary influenza symptoms and fever. The primary influenza symptoms included cough, sore throat, headache, nasal congestion, body aches and pains, and fatigue. Symptoms were considered alleviated when all were decreased to ≤1 and decrease persisted unchanged ≥ 21.5 hours. Fever was considered alleviated when maintained at < 38.0°C (age 20 to < 65 years) or < 37.8°C (age ≥ 65 years) ≥ 21.5 hours; Test type: Superiority or Other; p = .05, Gehan-Wilcoxon — A step-down approach was applied to the primary analysis, with the higher dose of favipiravir first tested against placebo

ADVERSE EVENTS:
Arm/Group | 1: Low Dose Favipiravir | 2: High Dose Favipiravir | Placebo
Serious Adverse Events (participants affected / at risk) | 2/132 | 0/189 | 1/197
Other Adverse Events (participants affected / at risk) | 47/132 | 65/189 | 79/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Low Dose Favipiravir (N=132) | 2: High Dose Favipiravir (N=189) | Placebo (N=197)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Patient experienced vulval abscess (CTCAE grade 3) on Day 9 of study. Treated with medication, event resolved 5 days later. Met seriousness criteria of hospitalization. Investigator considered event not related to study drug.
hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Patient experienced hepatic encephalopathy (CTCAE grade 1) on Day 4 of study. Treatment not required, event resolved 2 days later. PMH of cirrohsis. Event met seriousness criteria of prolonged hospitalization. Determined as unrelated to study drug.
bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Bronchial obstruction (CTCAE grade 1) Day 2 of study (placebo cohort). Withdrawn from study. Treated with medication, event resolved 4 days later. Met serious criteria of hospitalization. Investigator considered event unrelated to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Low Dose Favipiravir (N=132) | 2: High Dose Favipiravir (N=189) | Placebo (N=197)
bronchitis (Infections and infestations) | 0 (0) | 5 (5) | 2 (2)
dizziness (Nervous system disorders) | 2 (2) | 4 (4) | 6 (6)
headache (Nervous system disorders) | 3 (3) | 4 (4) | 9 (9)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2)
diarrhoea (Gastrointestinal disorders) | 3 (3) | 9 (9) | 10 (10)
nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 9 (9)
rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
proteinuria (Renal and urinary disorders) | 1 (1) | 4 (4) | 1 (1)
blood fibrinogen increased (Investigations) | 4 (4) | 3 (3) | 6 (6)
blood uric acid increased (Investigations) | 3 (3) | 7 (7) | 5 (5)
urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (4)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5)
alanine aminotransferase increase (Investigations) | 0 (0) | 3 (3) | 6 (6)
blood triglycerides increased (Investigations) | 2 (2) | 2 (2) | 4 (4)
INR increased (Investigations) | 0 (0) | 0 (0) | 5 (5)
ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
APTT prolonged (Investigations) | 0 (0) | 0 (0) | 3 (3)
aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
blood creatinine increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
WBC decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
neutrophil count increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
ketonuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
otitis media (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
tonsillits (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
pharyngitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
sinusitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
parasthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0)
tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
aphthous stomatitis (Gastrointestinal disorders) | 1 | 1 | 1
constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1)
pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 2 (2) | 3 (3)
gamma-glutamyl transferase increased (Investigations) | 0 (0) | 3 (3) | 3 (3)
lymphocyte count decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
bilibrubin urine (Investigations) | 0 (0) | 2 (2) | 0 (0)
hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
WBC increased (Investigations) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days